CLINICAL TRIAL: NCT06182150
Title: PAUSE-Cardio: Mitigating Depression, Anxiety, and Stress Among Women's Sport Student- Athletes Through a Moderate-Intensity Exercise Intervention
Brief Title: Mitigating Mental Health Issues Among Women's Sport Student-Athletes Through a Moderate-Intensity Exercise Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-0810
Record Dates: First submitted 2023-12-11; First posted 2023-12-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Depression; Anxiety; Stress, Psychological
Keywords: Exercise Intervention
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PAUSE-Cardio Moderate-Intensity Exercise Arm (Experimental): Arm receiving moderate-intensity indoor cycling exercise once weekly for 4 weeks.
  Interventions: Behavioral: Moderate-Intensity Indoor Cycling Exercise

INTERVENTIONS:
Behavioral: Moderate-Intensity Indoor Cycling Exercise — The 45-minute indoor cycling moderate-intensity cardiovascular exercise will take place once a week over four weeks. The group fitness-based class consists a 5-minute warm-up, a 35-minute conditioning segment, and a 5-minute cooldown.

SUMMARY:
The goal of this clinical trial is to learn about moderate-intensity indoor cycling interventions in women's sport student-athletes transitioning into college and collegiate sport. The main question[s] it aims to answer are:

Aim 1: Establish preliminary feasibility for the intervention based on recruitment and retention rates.

Aim 2: Assess efficacy through comparison of pre- and post-intervention mental health outcomes scores between experimental and control groups.

Exploratory Aim 3: Explore associations between exercise, athletic, and academic identities and mental health issues post-intervention.

Participants will complete an online questionnaire. This online questionnaire will be given before the program begins and after the 4 weeks. The questionnaire will ask about the participants' basic information, the participants' experience with exercise, and the participants' transition experience including mental, physical, and social factors.

Participants will be asked to attend an in-person 45-minute exercise class once a week at the University of North Carolina at Chapel Hill (UNC) Student Recreation Center.

Participants enrolled in the program will be asked to complete a self-report form during each weekly practice including heart rate (before and after practice) and ratings of perceived exertion. Heart rate will be measured during practice, smart devices (i.e., Apple Watch, FitBit) are not required.

DETAILED DESCRIPTION:
Purpose: The goal of this pilot study is to examine the relationship between mental health concerns (e.g., anxiety, depression, and stress) and PAUSE-Cardio, a 4-week moderate-intensity cardiovascular exercise intervention program for women's sport student-athletes transitioning into college and collegiate sport.

The investigators hypothesize that at least 70% of participants will be retained for the length of the intervention, including completion of the Qualtrics survey at T1 and T2. Additionally, the investigators hypothesize that symptoms of depression, anxiety, and stress will be significantly decreased post-intervention compared to pre-intervention following moderate-intensity exercise program completion.

Participants: Participants will consist of twenty-two women's sport student-athletes (N=22) ages 18 and older in the participants' first two years of undergraduate study. Participants must be actively practicing an intramural sport, club sport, varsity collegiate sport, or recreational sport.

Procedures: The study design will be a mixed-methods pilot study employing moderate-intensity cardiovascular exercise. Results will be assessed with a longitudinal self-report survey of valid and reliable psychometric measures and free response items. All measurements and questions will be compiled into one Qualtrics-based survey that will be administered two times (pre-program [T1] and post-program [T2]). Study-specific moderate-intensity exercise will be administered once weekly for four weeks in a group fitness setting for 45 minutes. The 45-minute class will consist of a 5-minute warm-up, a 35-minute conditioning segment, and a 5-minute cooldown. This multipart study is gathering data through a mixed-methods longitudinal design in conjunction with a prospective cohort design. Data collection is utilizing Qualtrics, an online survey platform, and administering PAUSE-Cardio, a 4-week moderate-intensity cardiovascular exercise intervention program. Individuals who are at least 18 years of age and self-identify as women's sport student-athletes within the participants' first two years of study in collegiate settings are invited to participate via social media, emails, flyers, and word of mouth. A self-report survey of valid and reliable psychometric quantitative measures and qualitative free-response items is being administered 4 weeks apart, pre-program (T1) and post-program (T2) to participants. The feasibility of the intervention program is being determined by examining recruitment and retention rates. To assess the preliminary efficacy of the intervention, within- and between-group comparisons are being conducted using aggregated data, including waitlist control data. In addition to the primary aims, an exploratory analysis is being conducted to investigate potential associations between exercise, athletic, and academic identities, and mental health issues.

ELIGIBILITY:
Inclusion Criteria:

* first- or second-year undergraduate student
* current participation in women's intramural sport, club sport, varsity collegiate sport, or recreational sport

Exclusion Criteria:

* individuals who did not meet the inclusion criteria
* those incapable of providing informed consent
* did not complete surveys at T1 and T2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Inclusion criteria include participants that self-identify as a women's sport student-athlete.
Enrollment: 5 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline in combined depression, stress, and anxiety symptomatology scores | Baseline, Week 4
  The Depression, Anxiety, and Stress Scale (DASS) utilizing 42 items on a 4-point Likert scale ranging from 0 to 3 (0=did not apply to me at all and 3=applied to me very much, or most of the time). Higher scores correlate with greater symptoms of depression, stress, and anxiety.

SECONDARY OUTCOMES:
Change from baseline in academic identity scores | Baseline, Week 4
  Academic Identity Measurement Scale, a 13-item measurement to investigate student identification with academics will be utilized. Each item will be scored on a 5-point Likert scale from 1 to 5 (1=strongly disagree and 5=strongly agree). Scores on the Academic Identity Measurement Scale were able to range from 13 to 65, with higher scores indicating greater identification with academics.
Change from baseline in athlete identity scores | Baseline, Week 4
  The Athlete Identity Measurement Scale (AIMS) was utilized to understand varying degrees of athletic identity within participants. AIMS is a reliable 10-item measure at the forefront of athletic identity measurement. Participants will be asked to complete 7 items from the AIMS, representing participant goals, friendships, and thoughts surrounding the sport the participant plays. The measurement was scored on a 7-point Likert scale (1=strongly disagree and 7=strongly agree) and scores are able to range from 7 to 35. Higher scores on the AIMS are suggestive of greater sports identity.
Change from baseline in exercise identity scores | Baseline, Week 4
  Participants responded to the full-form Exercise Identity Scale, a 9-item instrument used to measure one's identification with exercise as it related to the concept of self. Participants responded to the 9 items with a 7-point Likert scale (1=strongly disagree and 7=strongly agree) and scores were able to range from 9 to 45. Higher scores on the Exercise Identity Scale represented a greater identification with exercise in relation to one's concept of self.

CONTACTS AND LOCATIONS:
Overall Officials: Emily G Thomas, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Student Recreation Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson DF, Cychosz CM. Development of an exercise identity scale. Percept Mot Skills. 1994 Jun;78(3 Pt 1):747-51. doi: 10.1177/003151259407800313. PMID 8084685
- [Background] Lochbaum M, Cooper S, Limp S. The Athletic Identity Measurement Scale: A Systematic Review with Meta-Analysis from 1993 to 2021. Eur J Investig Health Psychol Educ. 2022 Sep 14;12(9):1391-1414. doi: 10.3390/ejihpe12090097. PMID 36135235
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Osborne, J. W. (1997). Identification with Academics and Academic Success among Community College Students. Community College Review, 25(1), 59-67.
- [Background] Qualtrics. (2013). Qualtrics (Version 37,892) [Computer software]. Provo, UT, USA